CLINICAL TRIAL: NCT00978263
Title: An Efficacy and Safety Comparison of Basal Insulin and OADs in Newly Diagnosed Type 2 Diabetes After Short-term Intensive Insulin Therapy
Brief Title: Comparison of Glargine and Oral Antidiabetic Drugs (OADs) in Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Department of Endocrinology, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChongqingMU
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Metformin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glargine (Experimental): Initial basal Insulin therapy was according to the dose administrated at bedtime in the last day hospitalization. basal Insulin doses were titrated every 3 days to achieve target FPG values between 80 and 130 mg/dl.
  Interventions: Drug: Glargine
- metformin-based Oral Antidiabetic Drugs (Experimental): Subject in metformin-based OAD group was visited every two weeks in the first month and the every four weeks for another five months. The subjects will start with Metformin 425mg bid, The dosage was titrated (up to 850mg bid) based on the fasting blood glucose every two weeks. If the patients fail to achieve the target, gliclazide-MR (Diamicron, Servier), or glimepiride (Amaryl, Sanofi-Aventis) would be added.
  Interventions: Drug: metformin-based Oral Antidiabetic Drugs

INTERVENTIONS:
Drug: metformin-based Oral Antidiabetic Drugs
  Other Names: Metformin and so on
  Arms: metformin-based Oral Antidiabetic Drugs
Drug: Glargine
  Other Names: Lantus
  Arms: Glargine

SUMMARY:
The investigators designed this prospective, randomized control study to compare the efficacy and safety between the basal insulin glargine therapy and metformin-based OADs after correction of the glucose toxicity with a short period of intensive insulin therapy.

DETAILED DESCRIPTION:
Detailed Description:

OBJECTIVE-Type 2 diabetes is associated with defects in insulin secretion and insulin sensitivity. Hyperglycemia may aggravate these defects, a feature known as glucose toxicity. Previous studies have shown that acute correction of hyperglycemia in subjects with long-standing type 2 diabetes gives only short-term improvement in glycemic control after discontinuation of insulin. The current study attempts to identify whether basal insulin glargine or metformin-based OADs for further management would have a long-term benefit in newly diagnosed type 2 diabetes after short-term intensive insulin therapy.

RESEARCH DESIGN AND METHODS-Newly diagnosed type 2 diabetic patients (fasting blood glucose >200 mg/dL or random blood glucose >300 mg/dL) will be hospitalized and treated with intensive insulin injection for 10 to 14 days. HbA1c were measured before intensive insulin injection. After discharge, patients will be randomized to receive basal insulin injection or metformin-based OADs for further management. Patients will be followed in our clinics and adjust their medication according to their blood glucose levels. HbA1c were measured 6 months later.After the six-month intervention, these patients were continually followed up for another six months. Subjects received an oral glucose tolerance test (OGTT) after the intensive insulin therapy and at the end of the 6th and 12th month.

EXPECTED RESULTS-We will expect that basal insulin glargine,compared with metformin-based OAD treatment,could more effectively maintain adequate glycemic control in newly diagnosed type 2 diabetes after short-term intensive insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed type 2 diabetic patients.
2. Drug naïve, with severe hyperglycemia (fasting plasma glucose>11.1mmol/L or random plasma glucose >16.7mmol/L)
3. Those who age between 30 and 70 years old and can inject insulin by themselves.

Exclusion Criteria:

1. Established type 1 diabetes or positive anti-glutamic acid decarboxylase antibody;
2. Malignancy, pregnancy or lactating;
3. History of ketoacidosis;
4. Hepatic dysfunction with alanine aminotransferase 2.5 times higher than the upper limit of normal; serum creatinine >2 mg/dl;
5. Poor blood pressure control (SBP>180mmHg or DBP >110mmHg);
6. Definite coronary artery disease, heart failure, left ventricular hypertrophy;
7. Severe anemia; acute or severe chronic diabetes complications;
8. BMI<18 kg/m2 or ≥41kg/m2;
9. History of alcohol abuse or drug abuse;
10. Mental disorder and other endocrine disorders; dysfunction of digestion and absorption;
11. Chronic diseases need long-term glucocorticoid treatment.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin (HbA1c) at month 6 | month 6
Change From Baseline in Glycosylated Hemoglobin at month 6 | Baseline and month 6

SECONDARY OUTCOMES:
Glycosylated Hemoglobin at month 12 | month 12
Change From Baseline in Glycosylated Hemoglobin at month 12 | Baseline and month 12
Number of Participants With Glycosylated Hemoglobin ≤ 7% | month 6
Number of Participants With Glycosylated Hemoglobin ≤ 7% | month 12
Number of Participants With Glycosylated Hemoglobin ≤ 6.5% | month 6
Number of Participants With Glycosylated Hemoglobin ≤ 6.5% | month 12
Fasting Plasma Glucose at week 2 | week 2
Fasting Plasma Glucose at week 4 | week 4
Fasting Plasma Glucose at week 8 | week 8
Fasting Plasma Glucose at week 12 | week 12
Fasting Plasma Glucose at week 16 | week 16
Fasting Plasma Glucose at week 20 | week 20
Fasting Plasma Glucose at week 24 | week 24
Fasting Plasma Glucose at week 32 | week 32
Fasting Plasma Glucose at week 40 | week 40
Fasting Plasma Glucose at week 48 | week 48
Homeostasis model assessment (HOMA)-β at month 6 | month 6
Insulinogenic index at month 6 | month 6
HOMA-IR at month 6 | month 6
Matsuda index at month 6 | month 6
Basal disposition index at month 6 | month 6
Early-phase disposition index at month 6 | month 6
Homeostasis model assessment (HOMA)-β at month 12 | month 12
Insulinogenic index at month 12 | month 12
HOMA-IR at month 12 | month 12
Matsuda index at month 12 | month 12
Basal disposition index at month 12 | month 12
Early-phase disposition index at month 12 | month 12
Diabetes Treatment Satisfaction Questionnaire status (DTSQs) version score | month 6
DTSQs score at month 12 | month 12
Audit of Diabetes Dependent Quality of Life (ADDQoL) score | month 6
ADDQoL score at month 12 | month 12
Cost at month 6 | month 6
Number of Participants with Hypoglycemia | up to 6 month
Number of hypoglycemia episodes | up to 6 month
Number of Participants with severe Hypoglycemia | up to 6 month
Number of severe hypoglycemia episodes | up to 6 month
Change From Baseline in Body Weight (month 6) | Baseline and month 6
Change From Baseline in Body Weight (month 12) | Baseline and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Principal Investigator — the First Affiliated Hospital, Chongqing Medical University, China
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China